CLINICAL TRIAL: NCT05298956
Title: Brain Substrates for Cardiovascular Stress Physiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Annie Ginty, Assistant Professor, Baylor University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1437574
Record Dates: First submitted 2022-02-21; First posted 2022-03-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Stress Reaction
MeSH Terms: conditions — Fractures, Stress | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): Participants will receive sham laser to the right forehead.
  Interventions: Other: Low-level laser therapy (LLLT)
- Transcranial infrared laser stimulation (Active Comparator): Participants will receive transcranial infrared laser stimulation to the right forehead.
  Interventions: Other: Low-level laser therapy (LLLT)

INTERVENTIONS:
Other: Low-level laser therapy (LLLT) — Sham Comparator: Participants will receive 8 counts of 60 seconds of the same laser to the right forehead, however the laser power will be turned off and will be 0 Watts.
  Transcranial infrared laser stimulation: Participants will receive 8 counts of 60 seconds of transcranial infrared laser stimulation to the right forehead. The wavelength will be 1064 nm and the laser power will be 3.4 Watts.

SUMMARY:
Transcranial infrared laser stimulation is a non-invasive neuromodulation technique. The study will examine the effect of transcranial infrared laser stimulation on cardiovascular and metabolic responses to stress.

DETAILED DESCRIPTION:
Physiological responses to stress may be a potential pathway by which psychological stress relates to cardiovascular disease. Disproportionate (metabolically exaggerated) stressor-evoked cardiovascular reactions may accelerate atherosclerosis or influence risk of greater cardiovascular disease endpoints. The aim of this project is to use an experimental approach to examine if neuromodulation (transcranial infrared laser stimulation) alters stressor-evoked metabolic and cardiovascular responses.

ELIGIBILITY:
Inclusion Criteria:

18-30 years old

Exclusion Criteria:

History of a diagnosed chronic medical or neurological disorder Current pregnancy Current illness or infection (e.g., cold, flu) Any condition that would prohibit them from engaging in physical exercise

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Oxygen consumption in response to acute psychological stress | Immediately following intervention (up to 60 minutes)
  This measurement takes into account oxygen consumption at baseline and during the stress task.
Heart rate in response to acute psychological stress | Immediately following intervention (up to 60 minutes)
  This measurement takes into account heart rate at baseline and during the stress task.
Additional heart rate in response to acute psychological stress | Immediately following intervention (up to 60 minutes)
  This measurement takes into account additional heart rate at baseline and during stress.

SECONDARY OUTCOMES:
Perceived stress | Immediately following intervention (up to 60 minutes)
  Ratings of perceived stressfulness (1 = not at all stressful, 7 = very stressful) of the acute psychological stress task

CONTACTS AND LOCATIONS:
Locations (1):
- Annie T. Ginty, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No